CLINICAL TRIAL: NCT04221256
Title: Dose-finding Study of Selective Serotonin Reuptake Inhibitors to Enhance Neuroplasticity
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closure due to COVID-19 pandemic
Sponsor: Burke Medical Research Institute (Other)
Responsible Party: Principal Investigator, Tomoko Kitago, Lab Director Human Motor Recovery Laboratory Assistant Professor, Burke Medical Research Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HMRL-002
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Stroke, Ischemic
Keywords: Selective Serotonin Reuptake Inhibitor; Neuroplasticity; Paired Associative Stimulation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: We propose a double-blinded, placebo-controlled crossover study to test a range of doses of escitalopram and a placebo control in enhancing PAS-induced plasticity in healthy individuals without neurological disease and patients with chronic stroke.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of SSRI (Experimental): Participants will be administered either 5, 10 or 20mg of SSRI escitalopram prior to paired associative stimulation.
  Interventions: Drug: Administration of SSRI escitalopram; Behavioral: Paired Associative stimulation
- Administration of Placebo (Placebo Comparator): Participants will be administered a placebo prior to paired associative stimulation
  Interventions: Behavioral: Paired Associative stimulation; Drug: Administration of Placebo

INTERVENTIONS:
Drug: Administration of SSRI escitalopram — Participants will be administered 5, 10 or 20mg of SRRI escitalopram prior to paired associative stimulation
  Arms: Administration of SSRI
Behavioral: Paired Associative stimulation — Participants will receive paired associative stimulation (transcranial magnetic stimulation and peripheral nerve stimulation) with an inter-stimulus interval length known to modulate corticospinal excitability.
Drug: Administration of Placebo — Participants will be administered a placebo prior to paired associative stimulation
  Arms: Administration of Placebo

SUMMARY:
The brain is able to change throughout life in response to learning, or injury, or to adapt to changes in the environment, which is known as neuroplasticity. Stroke survivors suffer disabling chronic motor impairments that have proven challenging to improve. Increasing neuroplasticity using selective serotonin reuptake inhibitors (SSRIs) is a promising approach to promote motor recovery in patients with stroke.

DETAILED DESCRIPTION:
The brain is able to change throughout life in response to learning, or injury, or to adapt to changes in the environment, which is known as neuroplasticity. Stroke survivors suffer disabling chronic motor impairments that have proven challenging to improve. Increasing neuroplasticity using selective serotonin reuptake inhibitors (SSRIs) is a promising approach to promote motor recovery in patients with stroke. Selective serotonin reuptake inhibitors (SSRIs) are currently widely used for treatment of depression, but they also have been shown to be able to enhance neuroplasticity. A single dose of SSRI has been shown to improve hand function in patients with chronic stroke. SSRIs also enhance neuroplasticity in healthy individuals, as shown using paired associative stimulation (PAS), a non-invasive method which causes the brain's excitability to change. However, the best dose of SSRI to increase neuroplasticity is not yet established.

The purpose of this study is to (1) find the effective dose of the SSRI escitalopram to modulate PAS-induced plasticity in patients with stroke and healthy individuals and (2) determine the variability of escitalopram's effect on PAS-induced plasticity between individuals. We measure neuroplasticity with PAS, which causes the brain's excitability to change. During PAS, you would receive electrical stimulation over your wrist and magnetic stimulation to their scalp (called transcranial magnetic stimulation, or TMS) to increase the excitability of the motor area of the brain. You will be asked to participate in a screening visit and 8 study visits separated by at least 1 week. At each study visit, you will be given a single dose of escitalopram (5, 10 or 20) or placebo, and we will measure your brain's change in excitability after PAS.

ELIGIBILITY:
Neurological Healthy Participants Inclusion criteria

1. Men and women aged 18 years and older.
2. Ability to give informed consent.

Exclusion criteria

1. Contraindications to TMS: epilepsy or other seizure history, ferromagnetic metallic implants in the head, or pacemaker
2. Current or history of neurological disorders or brain lesions such as stroke, multiple sclerosis, tumor, traumatic brain injury, spinal cord injury
3. Diagnosis of major depressive disorder or other psychiatric disorder
4. Currently taking escitalopram or another selective serotonin reuptake inhibitor
5. Currently taking or have taken in the past month other medications or supplements that have known interactions with escitalopram or can precipitate serotonin syndrome when taken in combination with escitalopram: monoamine oxidase inhibitors, methylene blue, linezolid, serotonin norepinephrine reuptake inhibitors (SNRI), triptans, tricyclic antidepressants (TCAs), fentanyl, lithium, tramadol, tryptophan, buspirone, amphetamines, St. John's wort
6. Known hypersensitivity to escitalopram or any of its inactive ingredients.
7. History of cerebral hemorrhage, gastrointestinal bleeding, or genitourinary bleeding.
8. History of prolonged QTc
9. Pregnant or breastfeeding
10. Social and/or personal circumstances that interfere with the ability to return for all study visits.

Stroke Patients Inclusion criteria

1. Men and women aged 18 years and older.
2. Ability to give informed consent.
3. History of ischemic stroke

Exclusion criteria

1. Contraindications to TMS: epilepsy or other seizure history, ferromagnetic metallic implants in the head, or pacemaker
2. Current or history of neurological disorders or brain lesions such as multiple sclerosis, tumor, traumatic brain injury, spinal cord injury
3. Diagnosis of major depressive disorder or other psychiatric disorder
4. Currently taking escitalopram or another selective serotonin reuptake inhibitor
5. Currently taking or have taken in the past month other medications or supplements that have known interactions with escitalopram or can precipitate serotonin syndrome when taken in combination with escitalopram: monoamine oxidase inhibitors, methylene blue, linezolid, serotonin norepinephrine reuptake inhibitors (SNRI), triptans, tricyclic antidepressants (TCAs), fentanyl, lithium, tramadol, tryptophan, buspirone, amphetamines, St. John's wort
6. Known hypersensitivity to escitalopram or any of its inactive ingredients.
7. History of cerebral hemorrhage, gastrointestinal bleeding, or genitourinary bleeding.
8. History of prolonged QTc
9. Pregnant or breastfeeding
10. Social and/or personal circumstances that interfere with the ability to return for all study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Change in motor evoked potential amplitude | Baseline, Up to 30 minutes Post PAS
  Assessment of corticospinal excitability

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Kitago, MD, Principal Investigator — Winifred Masterson Burke Medical Research Institute
Locations (1):
- Burke Neurological Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No